CLINICAL TRIAL: NCT05869643
Title: A Phase 2a, Randomized, Double-Blinded, Placebo-Controlled, Multicenter Study to Investigate the Antiviral Effect, Safety, Tolerability, and Pharmacokinetics of STP0404 in Adults With HIV-1 Infection
Brief Title: A Clinical Trial of STP0404 in Adults With HIV-1 Infection
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: ST Pharm Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STP-POC-001
Record Dates: First submitted 2023-04-17; First posted 2023-05-22 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: HIV-1-infection

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Initial randomization to Cohort 1 or 2 will not be blinded. However, randomization within each cohort to either receive STP0404 or matching placebo is blinded.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Cohort 1 STP0404 (Experimental)
  Interventions: Drug: Low-dose STP0404 (Pirmitegravir)
- Cohort 1 (Placebo Comparator)
  Interventions: Drug: Placebo
- Cohort 2 STP0404 (Experimental)
  Interventions: Drug: Medium-dose STP0404 (Pirmitegravir)
- Cohort 2 (Placebo Comparator)
  Interventions: Drug: Placebo
- Cohort 3 STP0404 (Experimental)
  Interventions: Drug: High-dose STP0404 (Pirmitegravir)
- Cohort 3 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Low-dose STP0404 (Pirmitegravir) — Once daily, oral capsule taken after breakfast
  Arms: Cohort 1 STP0404
Drug: Medium-dose STP0404 (Pirmitegravir) — Once daily, oral capsule taken after breakfast
  Arms: Cohort 2 STP0404
Drug: High-dose STP0404 (Pirmitegravir) — Once daily, oral capsule taken after breakfast
  Arms: Cohort 3 STP0404
Drug: Placebo — Matching placebo capsule, taken orally once daily after breakfast
  Arms: Cohort 1; Cohort 2; Cohort 3

SUMMARY:
The purpose of this study is to evaluate the antiviral effect, safety, tolerability, and pharmacokinetics of STP0404 in adult participants living with Human Immunodeficiency Virus Type 1 (HIV-1) infection.

ELIGIBILITY:
Inclusion Criteria:

* Have a confirmed HIV-1 infection in the documented medical record or at screening.
* Have never received any ARTs (i.e., treatment-naïve) before screening or only received one ARV regimen (2 or 3 drugs) at least 12 weeks before screening and/or received any monotherapy ≤10 days in a clinical trial setting at least 12 weeks before screening. Participants with a documented history of PrEP and/or PEP therapy but discontinued at least 8 weeks prior to screening are also eligible for inclusion.
* Have a CD4+ cell count ≥200 cells/mm3 at screening.

Exclusion Criteria:

* Have a hepatitis B surface antigen or positive hepatitis C virus antibody at screening. An HCV confirmation (HCV RNA test) will be performed at a central laboratory if the HCV antibodies screening result is positive. If the HCV RNA test result is negative, the participant will be eligible.
* Have a positive drug screen for amphetamines, barbiturates, cocaine, opiates, benzodiazepines, heroin, or phencyclidine. However, if in the opinion of the investigator, positive drug screen results may be due to prescription medication for therapeutic purposes (e.g., prescription Adderall for ADHD), eligibility decision shall rely on the investigator's medical judgment and should be documented.
* Have a history of regular alcohol consumption, defined as an average weekly intake of >14 drinks (males) or >7 drinks (females), within 6 months of screening and/or has positive alcohol screen at screening and baseline.
* Have received the following treatments as PrEP or PEP (≥1 dose) prior to screening: monoclonal antibodies, HIV-1 maturation inhibitors, and long-acting INSTIs (such as cabotegravir).
* Pregnant or lactating females.
* Have a history of clinically relevant pancreatitis or hepatitis within the previous 6 months.
* Participant received any allosteric HIV-1 integrase inhibitor (ALLINI, ≥1 dose) and/or received any long-acting ARVs (marketed or investigational, ≥1 dose) prior to screening.
* Have previously failed an INSTIs-containing regimen.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-05-23 (Actual); Primary Completion 2026-04-10 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
HIV-1 RNA copies change in plasma | Day 1, Day 11
  Change in plasma HIV-1 RNA log10 copies from baseline to Day 11 following a 10-day treatment period at each dose level.
Total Number of Adverse Events (AEs) occurring through Day 11 | Through day 11
  Cumulative number of AEs occurring from Day 1 through Day 11 at each dose level and placebo in treatment-naïve adults with HIV-1 infection, regardless of treatment discontinuation, and use of prohibited medications. The severity of the AE will be rated as per the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events Corrected Version 2.1, July 2017. These will be descriptively summarized.
Total Number of Serious Adverse Events (SAEs) occurring through Day 11 | Through day 11
  Cumulative number of SAEs occurring from Day 1 through Day 11 at each dose level and placebo in treatment-naïve adults with HIV-1 infection, regardless of treatment discontinuation, use of prohibited medications, and death are included in the endpoint. These will be descriptively summarized.
Mean area under the concentration-time curve from zero to 24 hours (AUC0-24h) | Day 1, Day 10
Mean observed maximum concentration after administration (Cmax) | Day 1, Day 10
Mean time to reach Cmax (Tmax) | Day 1, Day 10
Mean observed concentration at 24 hours after administration (C24h) | Day 2, Day 4, Day 7, Day10, Day 11
Mean area under the concentration-time curve to infinite time (AUCinf) | Day 10
Mean area under the concentration-time curve to time t (AUCt) | Day 10
Mean terminal half-life (t1/2) | Day 10
Mean apparent oral clearance (CL/F) | Day 10
Mean apparent volume of distribution (Vd/F) | Day 10

SECONDARY OUTCOMES:
HIV-1 RNA copies change in plasma from baseline to post-dose timepoints | Day 1, Day 2, Day 4, Day 7, Day 10, Day 11
HIV-1 RNA change in plasma from baseline to nadir over 11 days. | Day 1 pre-dose, Day 11
Plasma HIV-1 RNA rate of decline over 11 days | Day 1, Day 2, Day 4, Day 7, Day 10, Day 11
Number of participants with HIV-1 RNA <400 copies/mL | Day 1, Day 2, Day 4, Day 7, Day 10, Day 11
  descriptive statistics.
Number of participants with HIV-1 RNA <50 copies/mL | Day 1, Day 2, Day 4, Day 7, Day 10, Day 11
CD4+ cell count change | Day 1, Day 11
STP0404 exposure-efficacy relationship in plasma HIV-1 RNA copies / CD4+ cell count | Day 1, Day 11
Emergence of drug resistance mutations. | Screening, Day 1, Day 4, Day 7, Day 11

CONTACTS AND LOCATIONS:
Locations (13):
- United States (13):
  - Kaiser Permenente Los Angeles Medical Center, Los Angeles, California
  - Ruane Clinical Research, Inc., Los Angeles, California
  - Midway Immunology and Research Center, Ft. Pierce, Florida
  - Schiff Center for Liver Diseases/University of Miami, Miami, Florida
  - Orlando Immunology Center, Orlando, Florida
  - USF Health South Tampa Center for Advanced Healthcare, Tampa, Florida
  - Be Well Medical Center, Berkley, Michigan
  - Saint Michael's Medical Center, Newark, New Jersey
  - South Jersey Infectious Disease, Somers Point, New Jersey
  - North Shore University Hospital, Manhasset, New York
  - Atrium Health Wake Forest Baptist Medical Center - PPDS, Winston-Salem, North Carolina
  - St Hope Foundation, Inc, Bellaire, Texas
  - North Texas Infectious Diseases Consultants, P.A., Dallas, Texas

IPD SHARING:
Plan to Share IPD: No